CLINICAL TRIAL: NCT03497845
Title: Randomized, Double-Blinded, Phase 2 Study to Assess Safety and Immunogenicity of Homologous and Heterologous Prime-Boost Vaccination Strategies With Stockpiled Inactivated Monovalent Influenza A(H5) Vaccines Administered Intramuscularly With Either AS03 or MF59® as Adjuvant
Brief Title: Assess the Safety & Immunogenicity of Prime-Boost Vaccination Strategies Using H5Nx Virus Vaccine Adjuvanted With AS03 or MF59
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BP-I-16-005
Record Dates: First submitted 2018-03-13; First posted 2018-04-13 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Influenza A Virus, H5N1 Subtype
Keywords: vaccine; adjuvant; Influenza in Birds; MF59; AS03
MeSH Terms: conditions — Influenza in Birds | interventions — AS03 adjuvant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- a VN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant (Experimental): Single dose of Vietnam (VN) (H5N1) vaccine with AS03 Adjuvant (Dose 1 = Day 1), followed by single dose of gf/Washington (WA) (H5N8) vaccine with AS03 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: VN; Biological: gf/WA; Biological: AS03 adjuvant
- b IN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant (Experimental): Single dose of IN (H5N1) vaccine with AS03 Adjuvant (Dose 1 = Day 1), followed by single dose of gf/WA (H5N8) vaccine with AS03 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: IN; Biological: gf/WA; Biological: AS03 adjuvant
- c dk/BANG with AS03 Adjuvant, then gf/WA with AS03 Adjuvant (Experimental): Single dose of dk/Bangladesh (BANG) (H5N1) vaccine with AS03 Adjuvant (Dose 1 = Day 1), followed by single dose of gf/WA (H5N8) vaccine with AS03 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: dk/BANG; Biological: gf/WA; Biological: AS03 adjuvant
- d gf/WA with AS03 Adjuvant, then IN with AS03 Adjuvant (Experimental): Single dose of gf/WA (H5N8) vaccine with AS03 Adjuvant (Dose 1 = Day 1), followed by single dose of IN (H5N1) vaccine with AS03 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: IN; Biological: gf/WA; Biological: AS03 adjuvant
- e dk/BANG with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant (Experimental): Two doses of dk/BANG (H5N1) vaccine with AS03 Adjuvant (Dose1 = Day 1; Dose 2 = Day 22), followed by single dose of bhg/Qinghai Lake(QL) (H5N1) vaccine with AS03 Adjuvant (Day 142).
  Interventions: Biological: dk/BANG; Biological: bhg/QL; Biological: AS03 adjuvant
- f gf/WA with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant (Experimental): Two doses of gf/WA (H5N3) vaccine with AS03 Adjuvant (Dose 1 = Day 1; Dose 2 = Day 22), followed by single dose of bhg/QL (H5N1) vaccine with AS03 Adjuvant (Day 142)
  Interventions: Biological: gf/WA; Biological: bhg/QL; Biological: AS03 adjuvant
- g VN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant (Experimental): Single dose of VN (H5N1) vaccine with MF59 Adjuvant (Dose 1 = Day 1), followed by single dose of gf/WA (H5N8) vaccine with MF59 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: VN; Biological: gf/WA; Biological: MF59 adjuvant
- h IN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant (Experimental): Single dose of IN (H5N1) vaccine with MF59 Adjuvant (Dose 1 = Day 1), followed by single dose of gf/WA (H5N8) vaccine with MF59 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: IN; Biological: gf/WA; Biological: MF59 adjuvant
- i dk/BANG with MF59 Adjuvant, then gf/WA with MF59 Adjuvant (Experimental): Single dose of dk/BANG (H5N1) vaccine with MF59 Adjuvant (Dose 1 = Day 1), followed by single dose of gf/WA (H5N8) vaccine with MF59 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: dk/BANG; Biological: gf/WA; Biological: MF59 adjuvant
- j gf/WA with MF59 Adjuvant, then IN with MF59 Adjuvant (Experimental): Single dose of gf/WA (H5N8) vaccine with MF59 Adjuvant (Dose 1 = Day 1), followed by single dose of IN (H5N1) vaccine with MF59 Adjuvant (Dose 2 = Day 22).
  Interventions: Biological: IN; Biological: gf/WA; Biological: MF59 adjuvant
- k dk/BANG with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant (Experimental): Two doses of dk/BANG (H5N1) vaccine with MF59 Adjuvant (Dose 1 = Day 1; Dose 2 = Day 22); followed by single dose of bhg/QL (H5N1) vaccine with MF59 Adjuvant (Day 142).
  Interventions: Biological: dk/BANG; Biological: bhg/QL; Biological: MF59 adjuvant
- l gf/WA with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant (Experimental): Two doses of gf/WA (H5N8) vaccine with MF59 Adjuvant (Dose 1 = Day 1; Dose 2 = Day 22), followed by single dose of bhg/QL (H5N1) vaccine with MF59 Adjuvant (Day 142).
  Interventions: Biological: gf/WA; Biological: bhg/QL; Biological: MF59 adjuvant

INTERVENTIONS:
Biological: VN — 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  Other Names: A/Vietnam/1203/2004 vaccine antigen strain H5N1
  Arms: a VN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; g VN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant
Biological: IN — 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  Other Names: A/Indonesia/05/2005 vaccine antigen strain H5N1
  Arms: b IN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; d gf/WA with AS03 Adjuvant, then IN with AS03 Adjuvant; h IN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; j gf/WA with MF59 Adjuvant, then IN with MF59 Adjuvant
Biological: dk/BANG — 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  Other Names: A/duck/Bangladesh/19097/2013 vaccine antigen strain H5N1
  Arms: c dk/BANG with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; e dk/BANG with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant; i dk/BANG with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; k dk/BANG with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant
Biological: gf/WA — 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  Other Names: A/gyrfalcon/Washington/41088-6/2014 vaccine antigen strain H5N8
  Arms: a VN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; b IN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; c dk/BANG with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; d gf/WA with AS03 Adjuvant, then IN with AS03 Adjuvant; f gf/WA with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant; g VN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; h IN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; i dk/BANG with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; j gf/WA with MF59 Adjuvant, then IN with MF59 Adjuvant; l gf/WA with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant
Biological: bhg/QL — 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  Other Names: A/barheaded goose/Qinghai Lake/1A/2005 vaccine antigen strain H5N1
  Arms: e dk/BANG with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant; f gf/WA with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant; k dk/BANG with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant; l gf/WA with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant
Biological: AS03 adjuvant — 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  Arms: a VN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; b IN with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; c dk/BANG with AS03 Adjuvant, then gf/WA with AS03 Adjuvant; d gf/WA with AS03 Adjuvant, then IN with AS03 Adjuvant; e dk/BANG with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant; f gf/WA with AS03 Adjuvant, then bhg/QL with AS03 Adjuvant
Biological: MF59 adjuvant — 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  Arms: g VN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; h IN with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; i dk/BANG with MF59 Adjuvant, then gf/WA with MF59 Adjuvant; j gf/WA with MF59 Adjuvant, then IN with MF59 Adjuvant; k dk/BANG with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant; l gf/WA with MF59 Adjuvant, then bhg/QL with MF59 Adjuvant

SUMMARY:
The main purpose of this study is to assess the ability of H5 influenza virus vaccines and adjuvants present in the National Pre-Pandemic Influenza Vaccine Stockpile (NPIVS) to generate an immune response to homologous and to antigenically distant heterologous H5 influenza virus strains.

The study is designed to evaluate the safety and immunogenicity of vaccination strategies with homologous or antigenically distant heterologous H5 influenza virus vaccines administered with AS03 or MF59 adjuvant.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or nonpregnant female 18 to 49 years of age, inclusive, on Day 1 (first vaccination).
2. Will avoid nonstudy vaccinations until 21 days after the last vaccination.
3. Provides written informed consent prior to the initiation of any study-related procedures.
4. Has a stable health status, as established by physical examination, vital sign measurements, and medical history.
5. Has access to a consistent and reliable means of telephone contact, which may be in the home, workplace, or by personal mobile electronic device.
6. Is able to understand and comply with planned study procedures.
7. Lives a reasonable distance from the site to be able to travel to and from the site for follow-up visits and agrees to go to the site for evaluation in the case of an adverse event.
8. Agrees to stay in contact with the site for the duration of the study, has no current plans to move from the study area, and provides updated contact information as necessary.

Exclusion Criteria:

1. Has a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol-9, thimerosal, or chicken protein), or allergy to squalene-based adjuvants or has had severe reactions following previous immunizations with contemporary influenza virus vaccines.
2. A woman who has a positive urine pregnancy test prior to vaccination in this study or a woman who is breastfeeding.
3. A female of childbearing potential (a) who refuses to use an acceptable method of birth control (b) from Day 1 (first vaccination) to end-of-study visit and, if sexually active, who has not used a reliable birth control method for at least 2 months prior to Day 1 (first vaccination).

   1. Female of childbearing potential is defined as post-onset menarche and premenopausal female capable of becoming pregnant. This does not include females who meet any of the following conditions: menopausal >1 year, tubal ligation >1 year, bilateral salpingo-oophorectomy, or hysterectomy.
   2. Adequate contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label, for example: abstinence from penile-vaginal intercourse; oral contraceptives, either combined or progestogen alone; injectable progestogen; implants of etonogestrel or levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device or intrauterine system; male partner sterilization at least 6 months prior to the female Day 1 (first vaccination), and this male is the sole partner for that subject (The information on the male sterility can come from the site personnel's review of the subject's medical records or interview with the subject on her medical history); male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).
4. Is immunosuppressed as a result of an underlying illness or treatment, or anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months prior to Day 1 (first vaccination).
5. Has an active neoplastic disease or a history of any hematologic malignancy. A subject with superficial skin cancer who does not require intervention other than local excision is not excluded.
6. Has long-term use (≥14 consecutive days) of glucocorticoids including oral or parenteral prednisone or equivalent (>20 mg total dose per day) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within 1 month prior to screening. (Low-dose [≤800 mcg/day of beclomethasone dipropionate or equivalent] inhaled and topical steroids are allowed).
7. Has a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
8. Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
9. Has a neurological or psychiatric diagnosis, which, although stable, is judged by the investigator to render the potential subject unable or unlikely to comply with the protocol or to provide accurate safety reports.
10. Has received immunoglobulin or other blood product (with the exception of Rho[D] immune globulin) within the 3 months prior to Day 1 (first vaccination).
11. Has received any live vaccine within 4 weeks or inactivated vaccines within 2 weeks prior to Day 1 (first vaccination). This includes seasonal influenza vaccines.
12. Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses. This includes potentially immune-mediated medical conditions such as Guillain-Barré syndrome, narcolepsy, current or history of autoimmune or chronic inflammatory disease.
13. Has a first-degree relative with narcolepsy.
14. Has an acute illness, including body temperature greater than 100.4°F, at screening, immediately prior to each vaccination or, per subject report, within 3 days prior to each vaccination. Subjects with an acute illness can be rescheduled for a vaccination as long as the vaccination visit is within the visit window. Note that subjects may return for randomization following resolution of the acute illness as long as recruitment remains open and subjects are within 14 days of signing consent.
15. Has a Grade 2 or greater (by US Food and Drug Administration toxicity grade) safety laboratory value at screening.
16. Has received an experimental agent (vaccine, biologic, device, blood product, or medication) within 1 month prior to Day 1 (first vaccination) in this study or plans receipt of an experimental agent during the study period.
17. Is participating or plans to participate in another interventional clinical study (either active or follow-up phase) during the study period.
18. Has received an influenza H5 vaccine in the past or has a history of H5 influenza infection prior to enrollment.
19. Has known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
20. Has a history of alcohol or drug abuse within 5 years prior to Day 1 (first vaccination).
21. Has a body mass index >35 kg/m2.
22. Has any condition that would, in the opinion of the investigator, place him or her at an unacceptable risk of injury or render him or her unable to meet the requirements of the protocol (including site of injection reactogenicity assessments).
23. Is a first-degree relative of any person working on this study: site or sponsor.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 720 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Optimal Research, San Diego, California
  - Optimal Research, Peoria, Illinois
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Central Kentucky Research Associates Inc, Lexington, Kentucky
  - Optimal Research, Rockville, Maryland
  - Rochester Clinical Research, Inc, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant: Two doses of dk/BANG (H5N1) vaccine with MF59 Adjuvant (Dose 1 = Day 1; Dose 2 = Day 22), followed by single dose of bhg/QL (H5N1) vaccine with MF59 Adjuvant (Day 142).
  dk/BANG: 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  bhg/QL: 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  MF59 adjuvant: 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
Period: Overall Study
Arm/Group | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant
Started | 60 | 58 | 61 | 60 | 59 | 62 | 59 | 60 | 61 | 59 | 61 | 60
Completed (Groups A-D and G-J completed Day 142, Groups E, F, K, L completed Day 262.) | 55 (Day 142) | 45 (Day 142) | 50 (Day 142) | 50 (Day 142) | 38 (Day 262) | 44 (Day 262) | 51 (Day 142) | 50 (Day 142) | 47 (Day 142) | 53 (Day 142) | 46 (Day 262) | 38 (Day 262)
Not Completed | 5 | 13 | 11 | 10 | 21 | 18 | 8 | 10 | 14 | 6 | 15 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | Total
Number analyzed (Participants) | 60 | 58 | 61 | 60 | 59 | 62 | 59 | 60 | 61 | 59 | 61 | 60 | 720
Age, Customized [Count of Participants; unit: Participants]
  Age of Participants: 18-<30 years old | 23 | 23 | 26 | 26 | 24 | 21 | 24 | 18 | 34 | 18 | 22 | 25 | 284
  Age of Participants: 30-<40 years old | 17 | 15 | 23 | 17 | 21 | 17 | 15 | 22 | 13 | 26 | 14 | 19 | 219
  Age of Participants: 40-49 years old | 20 | 20 | 12 | 17 | 14 | 24 | 20 | 20 | 14 | 15 | 25 | 16 | 217
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 35 | 40 | 38 | 31 | 43 | 31 | 42 | 28 | 35 | 38 | 430
  Male | 23 | 26 | 26 | 20 | 21 | 31 | 16 | 29 | 19 | 31 | 26 | 22 | 290
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race of Participants: White | 51 | 42 | 42 | 49 | 42 | 47 | 44 | 48 | 45 | 41 | 42 | 42 | 535
  Race of Participants: Black or African American | 8 | 10 | 14 | 5 | 13 | 11 | 10 | 6 | 12 | 11 | 14 | 8 | 122
  Race of Participants: Asian | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 2 | 4 | 1 | 1 | 19
  Race of Participants: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Race of Participants: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race of Participants: Multiracial | 0 | 5 | 4 | 5 | 2 | 2 | 2 | 4 | 2 | 3 | 4 | 7 | 40
  Race of Participants: Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity of Participants: Hispanic or Latino | 4 | 7 | 6 | 5 | 6 | 5 | 7 | 7 | 5 | 4 | 7 | 5 | 68
  Ethnicity of Participants: Not Hispanic or Latino | 56 | 51 | 55 | 55 | 53 | 57 | 52 | 53 | 56 | 55 | 54 | 55 | 652
Body Mass Index (BMI) (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.637 (4.4123) | 26.750 (5.3287) | 27.561 (5.1079) | 26.840 (4.4868) | 26.458 (4.4476) | 26.495 (4.2461) | 26.798 (4.6794) | 27.297 (4.5460) | 26.457 (4.7881) | 26.824 (3.9945) | 26.867 (4.0300) | 26.268 (4.7620) | 26.771 (4.5691)

OUTCOME MEASURES:

1. Primary Outcome: Number of Local Adverse Reactions to 2-dose and 3-dose H5 Influenza Vaccination Series
Description: Safety of 2-dose and 3-dose H5 influenza vaccination series as determined by occurrence of mild, moderate, or severe solicited local reactogenicity symptoms.
  Subjects in A-D and G-J did not receive 3 doses
Time Frame: 8 days post-vaccination
Population: If a subject experienced multiple occurrences of the same solicited local AE, only the most severe solicited local AE was counted. If a subject had multiple AEs the number of events analyzed may be greater than the overall number of participants analyzed.
  Subjects in A-D and G-J did not receive 3 doses
Measure: Number; unit: Events
Arm/Group | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant
Number analyzed (Participants) | 60 | 58 | 61 | 60 | 59 | 62 | 59 | 60 | 61 | 59 | 61 | 60
Events
  AEs in subjects who received Dose 1 : Mild | 43 | 32 | 35 | 37 | 28 | 35 | 18 | 21 | 22 | 27 | 25 | 22
  AEs in subjects who received Dose 1 : Moderate | 3 | 5 | 6 | 4 | 3 | 10 | 1 | 0 | 1 | 2 | 2 | 1
  AEs in subjects who received Dose 1 : Severe | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs in subjects who received Dose 2 : Mild | 27 | 28 | 27 | 23 | 23 | 33 | 16 | 17 | 16 | 18 | 16 | 15
  AEs in subjects who received Dose 2 : Moderate | 5 | 4 | 3 | 3 | 5 | 3 | 0 | 0 | 4 | 2 | 2 | 3
  AEs in subjects who received Dose 2 : Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs in Subjects who received Dose 3 : Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 59 | 62 | 0 | 0 | 0 | 0 | 61 | 60
  AEs in Subjects who received Dose 3 : Mild |  |  |  |  | 17 | 17 |  |  |  |  | 10 | 6
  AEs in Subjects who received Dose 3 : Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 59 | 62 | 0 | 0 | 0 | 0 | 61 | 60
  AEs in Subjects who received Dose 3 : Moderate |  |  |  |  | 5 | 3 |  |  |  |  | 1 | 0
  AEs in Subjects who received Dose 3 : Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 59 | 62 | 0 | 0 | 0 | 0 | 61 | 60
  AEs in Subjects who received Dose 3 : Severe |  |  |  |  | 0 | 0 |  |  |  |  | 0 | 0

2. Primary Outcome: Number of Systemic Adverse Reactions to 2-dose and 3-dose H5 Influenza Vaccination Series
Description: Safety of 2-dose and 3-dose H5 influenza vaccination series as determined by occurrence of mild, moderate, or severe solicited systemic reactogenicity symptoms Subjects in A-D and G-J did not receive 3 doses
Time Frame: 8 days post-vaccination
Population: If a subject experienced multiple occurrences of the same solicited local AE, only the most severe solicited local AE was counted.
  Number Analyzed per Row = Participants with available data Subjects in A-D and G-J did not receive 3 doses
Measure: Number; unit: Events
Arm/Group | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant
Number analyzed (Participants) | 60 | 58 | 61 | 60 | 59 | 62 | 59 | 60 | 61 | 59 | 61 | 60
Events
  AEs in subjects who received dose 1 : Mild | 45 | 41 | 32 | 43 | 23 | 37 | 29 | 28 | 29 | 21 | 32 | 23
  AEs in subjects who received dose 1 : Moderate | 6 | 12 | 8 | 19 | 6 | 19 | 13 | 2 | 6 | 6 | 5 | 19
  AEs in subjects who received dose 1 : Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs in subjects who received dose 2 : Mild: number analyzed (Participants) | 57 | 54 | 58 | 56 | 52 | 58 | 55 | 56 | 56 | 54 | 59 | 51
  AEs in subjects who received dose 2 : Mild | 39 | 33 | 22 | 46 | 17 | 40 | 16 | 6 | 24 | 4 | 17 | 11
  AEs in subjects who received dose 2 : Moderate: number analyzed (Participants) | 57 | 54 | 58 | 56 | 52 | 58 | 55 | 56 | 56 | 54 | 59 | 51
  AEs in subjects who received dose 2 : Moderate | 19 | 10 | 7 | 20 | 8 | 21 | 4 | 0 | 3 | 6 | 6 | 2
  AEs in subjects who received dose 2 : Severe: number analyzed (Participants) | 57 | 54 | 58 | 56 | 52 | 58 | 55 | 56 | 56 | 54 | 59 | 51
  AEs in subjects who received dose 2 : Severe | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AEs in subjects who received dose 3 : Mild: number analyzed (Participants) | 0 | 0 | 0 | 0 | 42 | 47 | 0 | 0 | 0 | 0 | 48 | 40
  AEs in subjects who received dose 3 : Mild |  |  |  |  | 19 | 32 |  |  |  |  | 11 | 9
  AEs in subjects who received dose 3 : Moderate: number analyzed (Participants) | 0 | 0 | 0 | 0 | 42 | 47 | 0 | 0 | 0 | 0 | 48 | 40
  AEs in subjects who received dose 3 : Moderate |  |  |  |  | 19 | 12 |  |  |  |  | 2 | 0
  AEs in subjects who received dose 3 : Severe: number analyzed (Participants) | 0 | 0 | 0 | 0 | 42 | 47 | 0 | 0 | 0 | 0 | 48 | 40
  AEs in subjects who received dose 3 : Severe |  |  |  |  | 1 | 1 |  |  |  |  | 0 | 0

3. Primary Outcome: Percentage of Participants With Serum Hemagglutination Inhibition (HAI) Antibody Seroprotection Against Vaccine Strains Following 2-dose H5 Influenza Vaccination Series
Description: Serum hemagglutination inhibition (HAI) antibody seroprotection rate (SPR)
Time Frame: Day 43
Population: Seroprotection Rate by Strain (with 95% confidence interval) of HAI antibodies at Day 43 (21 days after Dose 2)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant: Two doses of dk/BANG (H5N1) vaccine with AS03 Adjuvant (Dose 1 = Day 1; Dose 2 = Day 22), followed by single dose of bhg/Qinghai Lake(QL) (H5N1) vaccine with AS03 Adjuvant (Day 142).
  dk/BANG: 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  bhg/QL: 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
  AS03 adjuvant: 0.5 mL vaccine (H5 vaccine antigen plus adjuvant) per dose
Arm/Group | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant
Number analyzed (Participants) | 53 | 52 | 54 | 52 | 40 | 45 | 51 | 52 | 51 | 51 | 46 | 38
percentage of participants
  A/gyrfalcon/Washington/41088-6/2014 (H5N8) (gf/WA) | 47.2 [33.7 to 60.6] | 40.4 [27.0 to 53.7] | 38.9 [25.9 to 51.9] | 50.0 [36.4 to 63.6] | 12.5 [2.3 to 22.7] | 80.0 [68.3 to 91.7] | 15.7 [5.7 to 25.7] | 15.4 [5.6 to 25.2] | 37.3 [24.0 to 50.5] | 11.8 [2.9 to 20.6] | 6.5 [0.0 to 13.7] | 63.2 [47.8 to 78.5]
  A/Indonesia/05/2005 (H5N1) (IN) | 13.2 [4.1 to 22.3] | 38.5 [25.0 to 51.7] | 11.1 [2.7 to 19.5] | 46.2 [32.6 to 59.7] | 32.5 [18.0 to 47.0] | 4.4 [0.0 to 10.5] | 0.0 [0.0 to 0.0] | 17.3 [7.0 to 27.6] | 3.9 [0.0 to 9.2] | 13.7 [4.3 to 23.2] | 10.9 [1.9 to 19.9] | 5.3 [0.0 to 12.4]
  A/duck/Bangladesh/19097/2013 (H5N1) (dk/BANG) | 26.4 [14.5 to 38.3] | 25.0 [13.2 to 36.8] | 31.5 [19.1 to 43.9] | 32.7 [19.9 to 45.4] | 67.5 [53.0 to 82.0] | 15.6 [5.0 to 26.1] | 3.9 [0.0 to 9.2] | 9.6 [1.6 to 17.6] | 33.3 [20.4 to 46.3] | 13.7 [4.3 to 23.2] | 50.0 [35.6 to 64.4] | 13.2 [2.4 to 23.9]
  A/Vietnam/1203/2004 (H5N1) (VN) | 75.5 [63.9 to 87.1] | 55.8 [42.3 to 69.3] | 44.4 [31.2 to 57.7] | 65.4 [52.5 to 78.3] | 37.5 [22.5 to 52.5] | 17.8 [6.6 to 28.9] | 39.2 [25.8 to 52.6] | 23.1 [11.6 to 34.5] | 33.3 [20.4 to 46.3] | 37.3 [24.0 to 50.5] | 26.1 [13.4 to 38.8] | 18.4 [6.1 to 30.7]
  A/barheaded goose/QinghaiLake/1A/2005(H5N1)bhg/QL | 28.3 [16.2 to 40.4] | 19.2 [8.5 to 29.9] | 20.4 [9.6 to 31.1] | 34.6 [21.7 to 47.5] | 22.5 [9.6 to 35.4] | 2.2 [0.0 to 6.5] | 13.7 [4.3 to 23.2] | 13.5 [4.2 to 22.7] | 9.8 [1.6 to 18.0] | 3.9 [0.0 to 9.2] | 6.5 [0.0 to 13.7] | 2.6 [0.0 to 7.7]

4. Primary Outcome: Percentage of Participants With Serum Hemagglutination Inhibition (HAI) Antibody Seroprotection Against Vaccine Strains Following 3-dose H5 Influenza Vaccination Series
Description: Serum hemagglutination inhibition (HAI) antibody seroprotection rate (SPR)
Time Frame: Day 163
Population: Seroprotection Rate by Strain (with 95% confidence interval) of HAI antibodies at Day 163 (21 days after Dose 3). Measurement of participants remaining rather than enrolled.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant
Number analyzed (Participants) | 40 | 45 | 46 | 38
percentage of participants
  A/gyrfalcon/Washington/41088-6/2014 (H5N8) (gf/WA) | 60.0 [44.8 to 75.2] | 82.2 [71.1 to 93.4] | 28.3 [15.2 to 41.4] | 52.6 [36.8 to 68.5]
  A/Indonesia/05/2005 (H5N1) (IN) | 75.0 [61.6 to 88.4] | 57.8 [43.3 to 72.2] | 50.0 [35.6 to 64.4] | 15.8 [4.2 to 27.4]
  A/duck/Bangladesh/19097/2013 (H5N1) (dk/BANG) | 90.0 [80.7 to 99.3] | 62.2 [48.1 to 76.4] | 63.0 [49.1 to 77.0] | 26.3 [12.3 to 40.3]
  A/Vietnam/1203/2004 (H5N1) (VN) | 90.0 [80.7 to 99.3] | 80.0 [68.3 to 91.7] | 63.0 [49.1 to 77.0] | 60.5 [45.0 to 76.1]
  A/barheaded goose/QinghaiLake/1A/2005(H5N1)bhg/QL | 72.5 [58.7 to 86.3] | 73.3 [60.4 to 86.3] | 45.7 [31.2 to 60.0] | 39.5 [23.9 to 55.0]

ADVERSE EVENTS:
Time Frame: 262 days
Description: Adverse events (AE) - If a subject experienced multiple occurrences of the same AE, only the most severe AE was counted
Arm/Group | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58 | 0/61 | 0/60 | 1/59 | 0/62 | 0/59 | 0/60 | 0/61 | 0/59 | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/58 | 1/61 | 0/60 | 2/59 | 0/62 | 2/59 | 1/60 | 0/61 | 0/59 | 4/61 | 1/60
Other Adverse Events (participants affected / at risk) | 46/60 | 45/58 | 44/61 | 43/60 | 47/59 | 47/62 | 40/59 | 36/60 | 40/61 | 41/59 | 45/61 | 42/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant (N=60) | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant (N=58) | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant (N=61) | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant (N=60) | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant (N=59) | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant (N=62) | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant (N=59) | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant (N=60) | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant (N=61) | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant (N=59) | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant (N=61) | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant (N=60)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major Depressive Episode with Suicidal Intent (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pregnancy with Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles/Ventricluar Premature Contractions (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankyloglossia, congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholin's Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | a VN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant (N=60) | b IN With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant (N=58) | c dk/BANG With AS03 Adjuvant, Then gf/WA With AS03 Adjuvant (N=61) | d gf/WA With AS03 Adjuvant, Then IN With AS03 Adjuvant (N=60) | e dk/BANG With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant (N=59) | f gf/WA With AS03 Adjuvant, Then Bhg/QL With AS03 Adjuvant (N=62) | g VN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant (N=59) | h IN With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant (N=60) | i dk/BANG With MF59 Adjuvant, Then gf/WA With MF59 Adjuvant (N=61) | j gf/WA With MF59 Adjuvant, Then IN With MF59 Adjuvant (N=59) | k dk/BANG With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant (N=61) | l gf/WA With MF59 Adjuvant, Then Bhg/QL With MF59 Adjuvant (N=60)
Injection site pain (General disorders) | 42 (42) | 35 (35) | 36 (36) | 35 (35) | 35 (35) | 36 (36) | 22 (22) | 26 (26) | 25 (25) | 28 (28) | 33 (33) | 25 (25)
Fatigue (General disorders) | 15 (15) | 14 (14) | 12 (12) | 14 (14) | 9 (9) | 16 (16) | 7 (7) | 6 (6) | 12 (12) | 8 (8) | 10 (10) | 6 (6)
Chills (General disorders) | 10 (10) | 7 (7) | 6 (6) | 12 (12) | 7 (7) | 14 (14) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Injection site swelling (General disorders) | 5 (5) | 2 (2) | 6 (6) | 3 (3) | 5 (5) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 5 (5) | 4 (4) | 5 (5) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 21 (21) | 16 (16) | 8 (8) | 17 (17) | 10 (10) | 22 (22) | 10 (10) | 11 (11) | 12 (12) | 7 (7) | 18 (18) | 11 (11)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 13 (13) | 14 (14) | 20 (20) | 13 (13) | 26 (26) | 8 (8) | 4 (4) | 14 (14) | 5 (5) | 11 (11) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 4 (4) | 4 (4) | 4 (4) | 10 (10) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 3
Nausea (Gastrointestinal disorders) | 9 (9) | 6 (6) | 7 (7) | 10 (10) | 10 (10) | 10 (10) | 5 (5) | 3 (3) | 3 (3) | 3 (3) | 5 (5) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 5 (5) | 7 (7) | 9 (9) | 9 (9) | 7 (7) | 3 (3) | 5 (5) | 5 (5) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03497845/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03497845/SAP_001.pdf